CLINICAL TRIAL: NCT05597943
Title: Randomized Control Trial to Investigate the Effect of a Smartphone Application for Gestational Diabetes Management on Postpartum Glucose Intolerance
Brief Title: mHealth Smartphone App and Postpartum Glucose Intolerance for Patients With GDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003186
Record Dates: First submitted 2022-10-17; First posted 2022-10-28 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Gestational Diabetes; PreDiabetes; Pregnancy Related; Pregnancy, High Risk
MeSH Terms: conditions — Diabetes, Gestational; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Malama Arm (Experimental): Participants enrolled in this arm will agree to using the Malama app to track glycemic management.
  Interventions: Behavioral: Malama App
- Control (No Intervention): Participants enrolled in this arm agree to standard management (FS log on phone, notebook, etc)

INTERVENTIONS:
Behavioral: Malama App — The Malama smartphone application is a gestational diabetes management app that syncs directly with commercially-available glucometers via Bluetooth, enabling both automatic blood glucose logging and providing interactive diet management/diet education tools. We aim to perform a pilot study assessing the impact of the Malama smartphone application on perinatal and postpartum outcomes in patients with GDM.
  Arms: Malama Arm

SUMMARY:
Without intervention, approximately 70% of women diagnosed with GDM will develop type 2 diabetes mellitus in their lifetime. Abnormal results of a 2 hour oral glucose tolerance test (OGTT) performed as early as 2 days postpartum are predictive of impaired glucose tolerance 1 year postpartum. The investigators hypothesize that use of the Malama smartphone application to optimize antenatal glycemic control will result in lower incidence of postpartum glucose intolerance, which may decrease long term risk of progression to diabetes mellitus.

DETAILED DESCRIPTION:
The effect of smartphone applications for gestational diabetes management on risk of postpartum glucose intolerance, antenatal glycemic control, and other perinatal outcomes is unknown.

This study is a randomized control trial in which patients diagnosed with gestational diabetes will be randomized to use of the Malama app vs. standard care as described above.

The primary aim of the study is to investigate if the incidence of postpartum glucose intolerance is lower in patients using the Malama app for gestational diabetes management compared to patients receiving standard care.

Secondary outcomes that will be investigated include several markers of maternal and neonatal perinatal morbidity. Maternal outcomes that will be investigated include postpartum hemoglobin A1c level, interval pregnancy weight gain, incidence of hypertensive disorders of pregnancy, cesarean delivery, operative delivery, postpartum hemorrhage, and advanced perineal lacerations. Neonatal secondary outcomes include gestational age at delivery, birthweight and incidence of large for gestational age infants, shoulder dystocia, NICU admission, length of NICU stay, neonatal blood glucose nadir, and need for neonatal IV glucose support.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women receiving prenatal, delivery, and postpartum care at Tufts Medical Center
2. Gestational diabetes diagnosed between 14 0/7 and 31 6/7 weeks gestation on basis of 1-hour glucose challenge test result of >=200 mg/dL or Carpenter-Coustan criteria
3. >= 18 years of age
4. Literate in English or Spanish (?additional languages pending app translation)
5. Access to or ownership of a smartphone compatible with Malama
6. Willing and able to sign the informed consent

Exclusion Criteria:

1. Unable to tolerate oral glucose tolerance test (i.e. history of gastric bypass surgery)
2. Diagnosis of pregestational diabetes
3. Prescribed medications for chronic disease that affect glucose metabolism (e.g., long term oral steroids)
4. Does not own smartphone compatible with Malama application
5. Severe life-limiting fetal anomaly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Malama app as intervention | 8-26 weeks
  The primary aim of the study is to investigate if the incidence of postpartum glucose intolerance is lower in patients using the Malama app for gestational diabetes management compared to patients receiving standard care.

SECONDARY OUTCOMES:
Postpartum hemoglobin A1c level | 6 months
  We will be measuring the postpartum A1c level to capture whether the mobile health app influences blood glucose levels based on glycemic control log method (app for intervention arm, pen-and-paper log for control).

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Z Ramos, MD, Study Director — Tufts Medical Center; Erika Werner, MD, MS, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No